CLINICAL TRIAL: NCT07001670
Title: The Effects of an 8-Week Tele-Yoga Program on Postoperative Recovery in Patients With Lung Cancer Undergoing Lung Resection
Brief Title: Investigation of the Effects of Tele-Yoga Training in Individuals With Lung Cancer Undergoing Lung Resection Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sevde Betül Kara, PhD Student, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-FTR-RK-01
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Period; Lung Cancer (Diagnosis)
Keywords: Exercise capacity; Pulmonary function; Muscle Strength; Dyspnea; Fatigue; Anxiety; Depression; Quality of Life; Exercise Therapy; Telemedicine; Rehabilitation
MeSH Terms: conditions — Lung Neoplasms; Disease; Dyspnea; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be performed by an investigator who is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Yoga Group (Experimental): Participants in this arm will receive an 8-week supervised tele-yoga program delivered via real-time video conferencing.
  Interventions: Other: Tele-Yoga Training
- Control Group (No Intervention): The control group will not receive any intervention.

INTERVENTIONS:
Other: Tele-Yoga Training — The Tele-yoga group will participate in real-time yoga sessions three times a week for eight weeks, including individual sessions for the first two weeks and small group sessions for the remaining six weeks, with all sessions supervised by a certified instructor. Each session will last approximately 45-60 minutes and include a 5-10 minute warm-up, 15-20 minutes of yoga postures, 15-20 minutes of yogic breathing exercises, and 5-10 minutes of relaxation and meditation.
  Arms: Tele-Yoga Group

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effects of an 8-week tele-yoga intervention in individuals with lung cancer who have undergone lung resection surgery. The intervention group will receive supervised yoga sessions via online synchronous video conferencing, while the control group will continue with standard post-operative care. The primary outcome is exercise capacity (6-minute walk test), with secondary outcomes including pulmonary function, respiratory and peripheral muscle strength, physical activity level, dyspnea, fatigue, sleep quality, anxiety and depression, and quality of life. It is hypothesized that tele-yoga will improve physical and psychological recovery post-surgery and may serve as a feasible home-based pulmonary rehabilitation alternative.

DETAILED DESCRIPTION:
Lung carcinoma, also referred to as pulmonary carcinoma, is a malignant tumor characterized by uncontrolled cell proliferation in the lung tissue, originating from epithelial cells. It is the most commonly diagnosed cancer type globally. Histopathologically, lung cancer is classified into two main categories: non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC). NSCLC constitutes approximately 85% of all lung cancer cases and is associated with high morbidity and mortality. According to the Tumor-Node-Metastasis (TNM) staging system developed by the American Joint Committee on Cancer (AJCC) and the Union for International Cancer Control (UICC), NSCLC is staged from I to IV. While SCLC has a lower prognostic value within the TNM system and is rarely operable, NSCLC is typically treated surgically in early stages.

Surgical treatment for early state of lung cancer includes lobectomy, pneumonectomy, segmentectomy, or wedge resection, depending on tumor location, lung function, and disease stage. The most commonly employed surgical approaches are thoracotomy, video-assisted thoracoscopic surgery (VATS), and robot-assisted thoracoscopic surgery (RATS). Although techniques such as VATS are associated with less postoperative pain, faster recovery, and better preservation of pulmonary function compared to thoracotomy, surgery still significantly reduces exercise capacity and contributes to long-term physical and psychological limitations.

Following lung resection, patients often experience a decline in exercise capacity, attributed to loss of lung parenchyma, ventilatory limitations, increased cardiac workload, thoracic pain, and muscle weakness. Dyspnea is prevalent in up to 60% of postoperative patients, many of whom did not experience dyspnea prior to surgery. Additionally, adjuvant chemotherapy and/or radiotherapy may cause pulmonary inflammation and fibrosis, further reducing lung function and quality of life. Sleep disturbances and psychological disorders such as anxiety and depression are also common during this period.

Exercise training is a non-pharmacological intervention that improves immune function and quality of life in cancer patients; however, traditional pulmonary rehabilitation programs are often underutilized postoperatively. There is increasing interest in mind-body exercise (MBE) modalities such as yoga, tai chi, and qigong, which integrate physical postures, breath control, and meditation. Among these, yoga has shown potential to improve exercise capacity, pulmonary function, muscle strength, fatigue, anxiety, depression, and sleep quality. Despite promising findings, there is a lack of evidence regarding the efficacy of structured yoga interventions specifically tailored for lung cancer patients post-surgery.

Furthermore, the transition from hospital to home poses challenges in ensuring the continuity and accessibility of rehabilitation services. Telehealth, defined as the provision of healthcare services via digital communication technologies, has emerged as a feasible platform for delivering home-based interventions. Tele-yoga, a form of remote supervised yoga practice, has shown benefits in various populations, including those with chronic obstructive pulmonary disease (COPD), heart failure, sleep apnea, and ankylosing spondylitis. However, no study has yet examined its application in post-surgical lung cancer patients.

Based on this gap in the literature, the present study aims to investigate the effects of an 8-week synchronized tele-yoga intervention on exercise capacity, pulmonary function, respiratory and peripheral muscle strength, physical activity level, dyspnea, fatigue, sleep quality, anxiety, depression, and health-related quality of life in patients who have undergone lung resection surgery for lung cancer. This will be the first randomized controlled trial to assess a comprehensive yoga-based telerehabilitation approach in this population. The findings may provide a cost-effective and practical home-based rehabilitation strategy to enhance physical and psychological recovery in lung cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years,
* Histologically confirmed diagnosis of Stage I-IIIA lung cancer according to the 9th edition of the AJCC Cancer Staging Manual,
* Underwent lobectomy, pneumonectomy, segmentectomy, or wedge resection via thoracotomy or video-assisted thoracoscopic surgery (VATS),
* An estimated life expectancy of ≥6 months,
* Karnofsky Performance Status score greater than 80% at study entry,
* Possession of the necessary equipment and access to a stable internet connection to enable participation in online interventions.

Exclusion Criteria:

* History of receiving radiotherapy or chemotherapy prior to surgery,
* Presence of severe dysfunction in vital organs such as the heart, brain, kidneys, or others,
* Having any comorbid condition that contraindicates participation in an exercise training program,
* Presence of serious postoperative complications,
* Cognitive impairments that hinder effective communication,
* Current participation in a structured and regular exercise program,
* Missing three consecutive weeks of sessions or completing less than 75% of the prescribed exercises,
* Voluntary withdrawal from the study by the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
The Six-Minute Walk Test (6MWT) | Change from Baseline at 8 weeks
  Distance walked in six minutes will be recorded. Test will be conducted according to the guideline of American Thoracic Society. Functional exercise capacity will be evaluated with the six-minute walk test. Patients will be walked in a 30-meter-long corridor for 6 minutes and the maximum walking distance will be measured. Before and after the test, heart rate, blood pressure and O2 saturation will be measured with pulse oximetry, and dyspnea and fatigue levels will be determined according to the Modified Borg scale.

SECONDARY OUTCOMES:
Incremental Shuttle Walk Test (ISWT) | Change from Baseline at 8 weeks
  The Incremental Shuttle Walk Test (ISWT) The Incremental Shuttle Walk Test adapted for chronic obstructive pulmonary disease (COPD) patients consists of 12 levels with progressively increasing walking speeds over a 10-meter course. The participant walks between two cones in response to auditory beeps from a laptop. The test continues until the participant is unable to maintain the required pace due to breathlessness or fatigue. The number of shuttles completed and total distance walked are recorded. VO₂max is calculated using the formula: VO₂max (ml/min/kg) = 4.19 + (0.025 × distance).
6-Minute Pegboard and Ring Test (6PBRT) | Change from Baseline at 8 weeks
  The 6PBRT evaluates upper extremity functional capacity by requiring participants to transfer rings from lower to upper pegs and back for 6 minutes. Participants may rest as needed, and the score is the total number of rings moved.
Pulmonary Function Tests (PFT) | Change from Baseline at 8 weeks
  Pulmonary function tests will be conducted using a portable spirometer, following the American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria.
Respiratory Muscle Strength Test (MIP/MEP) | Change from Baseline at 8 weeks
  Using a portable electronic oral pressure measurement device, maximal inspiratory pressure (MIP) and expiratory pressure (MEP) are measured per ATS/ERS recommendations. The highest value from three reproducible efforts is recorded in centimetres of water (cmH2O) and as a percentage of the expected value.
Peripheral Muscle Strength (Handgrip Strength Test) | Change from Baseline at 8 weeks
  Handgrip strength is measured using a dynamometer. Participants perform three trials with each hand, and the highest score is recorded in kg.
Physical Activity Level (IPAQ-SF) | Change from Baseline at 8 weeks
  Physical activity level is assessed using the Turkish-validated version of the International Physical Activity Questionnaire - Short Form (IPAQ-SF). This self-reported questionnaire evaluates physical activity performed in the last 7 days across different intensity levels (walking, moderate, and vigorous activity). Results are expressed in Metabolic Equivalent of Task (MET)-minutes/week.
  Scores range from 0 to an open-ended maximum depending on the amount and intensity of physical activity reported.
  Higher scores indicate a better outcome, reflecting a higher level of physical activity.
Dyspnea Assessment (Cancer Dyspnea Scale - CDS) | Change from Baseline at 8 weeks
  Dyspnea severity is measured using the validated Turkish version of the Cancer Dyspnea Scale (CDS). This self-reported scale evaluates dyspnea in cancer patients through three subscales: effort, discomfort, and anxiety related to breathing.
  The total CDS score ranges from 0 to 27, with each subscale consisting of items rated on a 4-point Likert scale (0-3).
  Higher scores indicate worse outcomes, reflecting greater severity of dyspnea and its associated components.
Fatigue Assessment (Fatigue Severity Scale - FSS) | Change from Baseline at 8 weeks
  Fatigue is assessed using the 9-item Fatigue Severity Scale, scored on a 7-point Likert scale. A mean score ≥4 indicates severe fatigue.
Sleep Quality (Pittsburgh Sleep Quality Index - PSQI) | Change from Baseline at 8 weeks
  Sleep quality is measured using the Pittsburgh Sleep Quality Index (PSQI), a validated self-reported questionnaire that assesses sleep quality over the past month. It includes seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
  The total PSQI score ranges from 0 to 21. Higher scores indicate worse sleep quality, with a score greater than 5 suggesting poor sleep quality.
Anxiety and Depression (Hospital Anxiety and Depression Scale - HADS) | Change from Baseline at 8 weeks
  Anxiety and depression are assessed using the HADS, with subscale cutoff scores of 10 for anxiety and 7 for depression.
Quality of Life (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30): | Change from Baseline at 8 weeks
  Cancer-specific quality of life is assessed using the validated Turkish version of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30). This instrument includes functional subscales (physical, role, emotional, cognitive, and social functioning), symptom subscales (e.g., fatigue, pain, nausea/vomiting), and a global health status/quality of life scale.
  Each item is scored on a Likert-type scale, and scores are linearly transformed to a 0-100 scale according to the EORTC scoring manual.
  For functional and global health status subscales, higher scores indicate better quality of life.
  For symptom subscales, higher scores indicate worse symptom burden.
Verbal Feedback | Post-intervention (Week 8)
  At the end of the 8-week intervention, participants in the intervention group will be asked to provide verbal feedback regarding safety, satisfaction, challenging poses, pros and cons of online sessions, and perceived effects of yoga.

CONTACTS AND LOCATIONS:
Overall Officials: Rengin Demir, Prof, Principal Investigator — Istanbul University - Cerrahpasa; Akif Turna, Prof, Principal Investigator — Istanbul University - Cerrahpasa; Sevde B Kara, PhD student, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Department of Thoracic Surgery, Cerrahpaşa Faculty of Medicine, Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No